CLINICAL TRIAL: NCT04240392
Title: Support Models for Addiction Related Treatment (SMART) Trial of Opioid Use Disorder OUD) in Pregnant Women
Brief Title: Treatment of Pregnant Women With OUD
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000027031; MAT-2018C2-12891 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2019-09-05; First posted 2020-01-27 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Opioid-use Disorder
Keywords: opioid; pregnant
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: This study will use a matched-pair cluster randomized trail design. The investigators will match clinical centers in pairs. The participants in each pair will be randomly assigned to either CC or ECHO using computer generated random numbers.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaborative Care (CC) (Experimental): The CC team includes an obstetrical provider and a nursing case manager. The obstetrician will see all participants, initially to discuss preferences for addiction treatment, buprenorphine, methadone (MAT) or no MAT. The obstetrician will see participants every 1-2 weeks, as needed and will provide prenatal care. The care team will meet at least monthly and review the participants' status. For research purposes, the CM will obtain informed consent, collect and enter results of the urine drug screen (UDS) into a database. At enrollment and at 26 and 34 weeks' gestation the care manager will ask participants to complete an assessment battery of self-reported measures.
  Interventions: Behavioral: Collaborative Care (CC)
- Extension for Community Healthcare Outcomes (ECHO) (Active Comparator): ECHO is a remote education model that provides mentorship and guided practice and participation in a learning community, via video conferencing. The practice members who participate in ECHO will include obstetricians and nurses as well as other members of the care team who wish to join. Providers are given access to a password-protected website containing the recorded sessions, a discussion board, and resource library. CME credits are available for each session and can motivate providers to attend.
  Interventions: Behavioral: Extension for Community Healthcare Outcomes (ECHO)

INTERVENTIONS:
Behavioral: Collaborative Care (CC) — The sites randomized to CC will have 4-6 on-site support visits at the outset of the study. These visits will occur during the first 3 months of the project. During these visits, study staff will again review buprenorphine induction procedures (heretofore referred to as "initiation" rather than "induction") and dosing of buprenorphine as well as therapeutic behavioral treatments. The investigators will provide the center with forms and educational materials as well as an "app" that can be run to help dosing during initiation procedures. At the same time, the investigators will teach obstetricians, nurses and support staff the principles of motivational interviewing. The investigators will set up visits for the CM to meet with a recovery coach trainer provided by the investigators' community partner.
  Arms: Collaborative Care (CC)
Behavioral: Extension for Community Healthcare Outcomes (ECHO) — The Weitzman Institute (WI), a community partner and provider for the ECHO condition, is a research and innovation center focused on improving care for medically underserved and special populations. Since 2013, CHCI/WI has provided education and technical assistance through an established video conference and online learning platforms to over 800 primary care providers and over 200 care team members who treat patients with chronic pain and opioid addiction. WI partners with national experts in pain care, substance abuse disorder, and MAT to create and deliver a robust training program for clinicians across the country through Project ECHO ®. The WI will work with the study team to develop and staff the sessions.
  Arms: Extension for Community Healthcare Outcomes (ECHO)

SUMMARY:
The investigators are testing two models of support for pregnant women with an opioid use disorder (OUD)

DETAILED DESCRIPTION:
The investigators are proposing a cluster randomized clinical trial to compare the effectiveness of two models of support for reproductive health clinicians to provide care for pregnant and postpartum women with an OUD: 1) a collaborative care (CC) approach based upon the Massachusetts Office-Based-Opioid Treatment (OBOT) Model that would provide onsite training, and support to providers and participants through the use of care managers (CMs) vs 2) a telesupport approach modeled on the Project Extension for Community Healthcare Outcomes (ECHO), a remote education model that provides mentorship and guided practice and participation in a learning community, via video conferencing.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Females age 18 or older
* Documented pregnancy in the medical record at less than 34 weeks gestation
* Delivery date no later than July 1, 2024
* Willingness to adhere to the study schedule
* Confirmed opioid use disorder by the DSM-5 Opioid Use Disorder questionnaire
* Ability to communicate in English
* No current plan to move out of the obstetrical provider treatment area within the study timeframe of approximately 44 weeks

Exclusion Criteria:

* Experiencing cognitive or emotional impairment that precludes the participant from providing informed consent
* Current hospitalization, incarceration, or institutionalization (if women present for care after institutionalization, participation is possible
* Current court case pending that would make incarceration likely during the study treatment period (approximately 44 weeks)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women with opioid use disorder
Enrollment: 230 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariadna Forray, MD, Principal Investigator — Yale University
Locations (11):
- United States (11):
  - Hartford Hospital, Hartford, Connecticut
  - Hospital of Central CT, New Britain, Connecticut
  - Yale New Haven Hospital Maternal Fetal Medicine Unit, New Haven, Connecticut
  - Yale New Haven Hospital Women's Center/Hill Health Center, New Haven, Connecticut
  - Coastal ObGyn & Midwifery, New London, Connecticut
  - OB Gyn Services PC, Norwich, Connecticut
  - Essex County ObGyn, Beverly, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - AFA Obstetrics & Gynecology, Concord, Massachusetts
  - Women's Health, Lowell General Hospital, Lowell, Massachusetts
  - Wesson's Women's Clinic UMASS Baystate, Springfield, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
De-Identified data will be made available to other researchers upon request. Please contact Dr. Yonkers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 years after the end of the study
Access Criteria: we will ask people to complete a request form

REFERENCES:
- [Derived] Kaufman JS, Yonkers KA, Maltz C, Friedhoff CM, Londono Tobon A, Mele A, Tessier-Kay M, Grechukhina O, Lipkind H, Byatt N, Forray A. Reporting Perinatal Substance Use to Child Protective Services: Obstetric Provider Perspectives on the Impact on Care. J Womens Health (Larchmt). 2024 Nov;33(11):1501-1508. doi: 10.1089/jwh.2023.0822. Epub 2024 May 21. PMID 38770764
- [Derived] Forray A, Mele A, Byatt N, Londono Tobon A, Gilstad-Hayden K, Hunkle K, Hong S, Lipkind H, Fiellin DA, Callaghan K, Yonkers KA. Support Models for Addiction Related Treatment (SMART) for pregnant women: Study protocol of a cluster randomized trial of two treatment models for opioid use disorder in prenatal clinics. PLoS One. 2022 Jan 13;17(1):e0261751. doi: 10.1371/journal.pone.0261751. eCollection 2022. PMID 35025898

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of participants occurred at one of the participating clinical sites. Clinical sites, not participants, were randomized to either CC or ECHO; therefore, all participants recruited from the same clinical site were randomized to the same model, CC or ECHO.
Pre-assignment Details: 230 pregnant participants were enrolled; however, two participants had their pregnancies end before they could engage in the intervention. Therefore, only 228 participants underwent the intervention.
Units Other Than Participants: clinical site
Groups:
- Collaborative Care (CC): The CC team includes an obstetrical provider and a nursing case manager. The obstetrician will see all participants, initially to discuss preferences for addiction treatment, buprenorphine, methadone (MAT) or no MAT. The obstetrician will see participants every 1-2 weeks, as needed and will provide prenatal care. The care team will meet at least monthly and review the participants' status. For research purposes, the CM will obtain informed consent, collect and enter results of the urine drug screen (UDS) into a database. At enrollment and at 26 and 34 weeks' gestation participants will complete an assessment battery of self-reported measures.
  Collaborative Care (CC): The sites randomized to CC will have 4-6 on-site support visits at the outset of the study. These visits will occur during the first 3 months of the project. During these visits, study staff will again review buprenorphine induction procedures (heretofore referred to as "initiation" rather than "induction") and dosing of buprenorphine as well as therapeutic behavioral treatments. The investigators will provide the center with forms and educational materials as well as an "app" that can be run to help dosing during initiation procedures. At the same time, the investigators will teach obstetricians, nurses and support staff the principles of motivational interviewing. The investigators will set up visits for the CM to meet with a recovery coach trainer provided by the investigators' community partner.
Period: Overall Study
Arm/Group | Collaborative Care (CC) | Extension for Community Healthcare Outcomes (ECHO)
Started | 126; 6 clinical site | 102; 6 clinical site
Completed Baseline | 113; 6 clinical site | 90; 6 clinical site
Completed Week 26 | 102; 6 clinical site | 81; 6 clinical site
Completed Week 36 | 96; 6 clinical site | 77; 6 clinical site
Completed 3 Month Postpartum | 102; 6 clinical site | 86; 6 clinical site
Completed | 102; 6 clinical site | 86; 6 clinical site
Not Completed | 24; 0 clinical site | 16; 0 clinical site
Not completed — Withdrawal by Subject | 13 | 4
Not completed — Lost to Follow-up | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Collaborative Care (CC) | Extension for Community Healthcare Outcomes (ECHO) | Total
Number analyzed (Participants) | 126 | 102 | 228
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (4.5) | 31.0 (4.9) | 31.4 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 102 | 228
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 20 | 38
  Not Hispanic or Latino | 102 | 80 | 182
  Unknown or Not Reported | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 6 | 16
  White | 98 | 77 | 175
  More than one race | 2 | 7 | 9
  Unknown or Not Reported | 14 | 12 | 26
Region of Enrollment [Number; unit: participants]
  United States | 126 | 102 | 228

OUTCOME MEASURES:

1. Primary Outcome: Treatment Engagement
Description: Dichotomous - A participant completes engagement if the baseline assessment is completed and the participant has had greater than 2 visits for treatment of OUD
Time Frame: 30 days from baseline
Population: The engagement cohort included individuals who did not enroll in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Collaborative Care (CC) | Extension for Community Healthcare Outcomes (ECHO)
Number analyzed (Participants) | 187 | 156
Participants
  Not engaged | 78 | 64
  Engaged | 109 | 92
Statistical Analysis 1: Comparison: Collaborative Care (CC) vs Extension for Community Healthcare Outcomes (ECHO); Test type: Superiority; p = 0.5340, Mixed Models Analysis; Generalized Linear Mixed Model; Odds Ratio (OR) = 1.369, 95% CI 2-sided [0.462 to 4.055]

2. Primary Outcome: Treatment Retention
Description: Dichotomous- A participant is considered to have been successfully retained in the study if the participant remained in treatment with no stoppage of greater than 1 month.
  The numbers reported below for 3 months postpartum differ from those in the Participant Flow, as the numbers in the Participant Flow represent only completed REDCap survey assessments. For the retention outcome, we could utilize additional sources of data collection, such as medical records, site reports, and treatment utilization forms (which were done more frequently than survey assessments), thus resulting in a higher N for this outcome.
Time Frame: delivery and three-month post-partum
Population: Data presented here is from all participants who completed assessments at each time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Collaborative Care (CC) | Extension for Community Healthcare Outcomes (ECHO)
Number analyzed (Participants) | 126 | 102
Participants
  Delivery: number analyzed (Participants) | 116 | 99
  Delivery: Not retained | 17 | 12
  Delivery: Retained | 99 | 87
  3 months post partum: number analyzed (Participants) | 114 | 95
  3 months post partum: Not retained | 18 | 11
  3 months post partum: Retained | 96 | 84
Statistical Analysis 1: Comparison: Collaborative Care (CC) vs Extension for Community Healthcare Outcomes (ECHO); At delivery; Test type: Superiority; p = 0.600, Mixed Models Analysis; Generalized Linear Mixed Model; Odds Ratio (OR) = 0.803, 95% CI 2-sided [0.326 to 1.979]
Statistical Analysis 2: Comparison: Collaborative Care (CC) vs Extension for Community Healthcare Outcomes (ECHO); At 3 months post partum; Test type: Superiority; p = 0.471, Mixed Models Analysis; Generalized Linear Mixed Model; Odds Ratio (OR) = 0.709, 95% CI 2-sided [0.254 to 1.975]

3. Primary Outcome: Patient Activation Measure (PAM)
Description: The PAM is a patient-centered questionnaire that measures health care knowledge, beliefs, skills and confidence in managing illnesses. The PAM has 13 items with a 5-point Likert response scale. The raw scores are summed and transformed to 0-100 metric (0 = lowest activation level, 100 = highest).
  The Week 26 numbers below are lower than those in the Participant Flow because participants were allowed to enter the study after 26 weeks of pregnancy and did not have a separate baseline and Week 26 PAM assessment; instead, it was counted as their baseline PAM assessment only. However, other study assessments were unique to week 26 and were completed concurrently with baseline assessments, which were counted separately, accounting for the higher N for Week 26 in the Participant Flow.
  The postpartum ECHO sample size is 85 rather than 86 because one participant skipped the PAM questions during their 3-month postpartum assessment.
Time Frame: baseline, week 26, week 36 and 3-monhts post-partum
Population: Data presented here is from all participants who completed assessments at each time frame.
  The numbers 117 and 94 represent the total number of participants with a PAM score recorded at any time point, as they were included in the analysis model. There were 17 participants who did not complete the PAM assessment at any time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Collaborative Care (CC) | Extension for Community Healthcare Outcomes (ECHO)
Number analyzed (Participants) | 117 | 94
score on a scale
  Baseline: number analyzed (Participants) | 113 | 90
  Baseline | 74.77 (19.03) | 76.6 (17.75)
  Week 26: number analyzed (Participants) | 51 | 49
  Week 26 | 78.32 (17.77) | 78.14 (18.11)
  Week 36: number analyzed (Participants) | 96 | 77
  Week 36 | 77.37 (16.35) | 78.55 (17.47)
  3 months post partum: number analyzed (Participants) | 102 | 85
  3 months post partum | 76.62 (17.26) | 78.25 (16.52)
Statistical Analysis 1: Comparison: Collaborative Care (CC) vs Extension for Community Healthcare Outcomes (ECHO); At week 36; Test type: Superiority; p = 0.518, Mixed Models Analysis; Repeated Measures Linear Mixed Model; Beta-coefficient = 1.53, 95% CI 2-sided [-3.13 to 6.19] — Beta-coefficient for treatment for time interaction term
Statistical Analysis 2: Comparison: Collaborative Care (CC) vs Extension for Community Healthcare Outcomes (ECHO); At 3 months post partum; Test type: Superiority; p = 0.893, Mixed Models Analysis; Repeated Measures Linear Mixed Model; Beta-coefficient = 0.32, 95% CI 2-sided [-4.41 to 5.06] — Beta-coefficient for treatment for time interaction term

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Collaborative Care (CC) | Extension for Community Healthcare Outcomes (ECHO)
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/102
Serious Adverse Events (participants affected / at risk) | 22/126 | 18/102
Other Adverse Events (participants affected / at risk) | 0/126 | 0/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Collaborative Care (CC) (N=126) | Extension for Community Healthcare Outcomes (ECHO) (N=102)
Hospitalization for opioid withdrawal (General disorders) | 4 | 0
Drug overdose (General disorders) | 2 | 2
Residential treatment admission (General disorders) | 1 | 3
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 13 | 10
Short Cervix effecting pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Fetal demise (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Thrombotic stroke (Cardiac disorders) | 0 | 1
Necrotizing Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT04240392/Prot_SAP_000.pdf